CLINICAL TRIAL: NCT03837912
Title: Intervention Based on the Use of Patient Feedback Collected for Improving Patient Safety in Spanish Primary Care (PC) Centres
Brief Title: Improving Patient Safety in Spanish Primary Care (PC) Centres
Acronym: SinergiAPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fundació d'investigació Sanitària de les Illes Balears (Other Government)
Collaborators: Ministerio de Economía y Competitividad, Spain (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CP17/00017
Record Dates: First submitted 2019-01-10; First posted 2019-02-12 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2020-03

CONDITIONS: Patient Safety
Keywords: cluster randomized controlled trial; primary health care; patient safety; patient-centred care; patient-reported experiences and outcomes measures; audit and feedback interventions.

STUDY DESIGN:
Intervention Model Description: Multi-centre, 12 month, two-arm, two-level cluster randomized controls trial (Primary Care professionals within Primary Care centres, with randomization at the centre level in a 1:1 ratio)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient reported safety experiences fed back to PC providers (Experimental): The intervention will consist in gathering patient-reported experiences and outcomes of the safety of the healthcare patients received in their PC centres during the previous 12 months. This information will be processed and fed back to their healthcare professionals to help them identify potential safety problems, and then target improvements based on problematic areas.
  Interventions: Behavioral: Patient reported safety experiences fed back to PC providers
- Patient reported safety experiences not fed back to providers (No Intervention): Waiting list: the practices allocated to the control group will receive the intervention (feedback report) after the trial finished (i.e., after post-intervention data collection has been completed).

INTERVENTIONS:
Behavioral: Patient reported safety experiences fed back to PC providers — The intervention will involve three key stages: a) Measurement: Patients will be invited to complete the Patient Reported Experiences and Outcomes of Safety in Primary Care (PREOS-PC) questionnaire using a tablet-computer. b) Feedback: Using a bespoke online tool, the information will be processed and presented to each centre in the form of a Feedback Report, which will offer comparisons with other centres along with a set of recommendations for addressing the problems identified. c) Action planning and change: centres will form an Action Planning Team, which will be responsible for analyzing the report, considering which area(s) should be improved, and developing, implementing and monitoring an action plan to address the safety problems identified.
  Arms: Patient reported safety experiences fed back to PC providers

SUMMARY:
Background:

Patient safety has been defined as "the avoidance, prevention, and amelioration of adverse outcomes or injuries stemming from the processes of healthcare"[1]. It has been on the research agenda for more than two decades, but more prominently since the report 'To Err is Human'[2]. To date concern about the safety of patients in hospital settings has driven most research in the field, and the knowledge about patient safety in the primary care (PC) setting is still sparse.

More emphasis on research on PC patient safety is needed because many safety incidents identified in hospitals actually originate in PC centres[3], which is where the overwhelming majority of healthcare is delivered[4]. That is especially in Spain, country with the highest PC frequentation figures in Europe, (average of 9.5 PC consultations per person per year[5]).

The overall aim of this study is to develop and evaluate an intervention targeted at PC professionals to improve patient safety in PC centres by providing them with feedback on patient perceptions, experiences and outcomes of patient safety.

Specific objectives:

1. To translate, cross-culturally adapt and validate the "Patient Reported Experiences and Outcomes of Safety in Primary Care" (PREOS-PC) instrument into the Spanish context.
2. To develop a feasible, acceptable, low-cost and scalable theory-based intervention targeted at PC professionals to improve patient safety in PC centres by providing them with feedback on patient perceptions, experiences, and outcomes of patient safety collected through the Spanish version of PREOS-PC.
3. To evaluate the acceptability and perceived utility of the intervention, and its effectiveness in improving safety climate, patient-reported patient safety, and reducing avoidable hospitalizations, when compared to usual care.

Method/design:

This study will involve 3 stages: Stage 1 (intervention development) will involve: a) qualitative study with end-users (PC providers) to explore the acceptability and utility of the proposed intervention, and potential implementation barriers; b) translation, cross-cultural adaptation and validation of the PREOS-PC survey for use in the Spanish context; c) development of the intervention components (feedback report and educational materials), and; d) development of an online tool to electronically administrate the PREOS-PC and to automatically generate and send feedback reports to PC centres. Stage 2 (piloting the intervention) will involve a feasibility study in 10 PC centres to inform refinement of the intervention and trial procedures. Stage 3 (evaluating the intervention) will involve: a) a cluster Randomized Controlled Trial to evaluate the impact of the intervention on patient safety culture, patient-reported safety experiences and outcomes, and avoidable hospital admissions, and; b) a qualitative study with PC providers to evaluate the acceptability and perceived utility of the intervention

DETAILED DESCRIPTION:
METHODS Description of the intervention The intervention will consist in gathering patient-reported experiences and outcomes of the safety of the healthcare patients received in their PC centres during the previous 12 months. This information will be processed and fed back to their PC professionals to help them identify potential problems, and then target improvements based on problematic areas.

The 3 stages of the intervention are:

1. Measurement: Patients will be approached in the waiting room, the study explained, and informed consent taken. The PREOS-PC questionnaire will be completed using a tablet-computer. Patients will be given a choice of whether they would prefer to self-complete the questionnaire or have it facilitated by the researcher.
2. Feedback: Using a bespoke online tool, the information for each PC centre will be collated and presented to the centres in the form of an automatically generated "Feedback Report", which will offer comparisons with other centres and also include a set of recommendations about how the problems identified could be addressed.
3. Action planning and change: Participating PC centres will form an Action Planning Team. Each team will comprise around four people working in the centres. The team will be responsible for receiving the Feedback Report, considering which area(s) should be targeted, and developing, implementing and monitoring an action plan for safety improvement.

This intervention is based on the Feedback Intervention Theory (FIT), which states that behaviour is regulated through comparison with standards or goals, and that feedback can draw attention to existing gaps[6]. FIT further postulates that once the gap has been identified, different methods can be followed in order to decrease it and attain the standard, including increasing the effort currently done[6], and implementing new strategies to address the problems identified. This could result in improving proximal outcomes (such as safety climate), and potentially impact more distal outcomes (e.g. incidence of safety events or avoidable hospitalizations).

Development and evaluation of the intervention The methods described below are based on the Medical Research Council guidance for the development and evaluation of complex interventions[7]. The development and evaluation of the intervention described above will involve three stages. Stage 1 (intervention development) will involve: a) a qualitative study with end-users (PC providers) to explore the acceptability and utility of the proposed intervention, and potential implementation barriers; b) translation, cross-cultural adaptation and validation of the PREOS-PC survey for use in the Spanish context; c) development of the intervention components (feedback report and educational materials), and; d) development of an online tool to administrate the PREOS-PC and to automatically generate and send feedback reports to PC centres. Stage 2 (piloting the intervention) will involve a feasibility study in 10 PC centres (260 professionals and 500 patients). Stage 3 (evaluating the intervention) will involve: a) a cluster randomized controlled trial (48 PC centres, 1248 professionals and 3600 patients) to evaluate the impact of the intervention on patient safety culture, patient-reported safety experiences and outcomes, and avoidable hospital admissions, and; b) a qualitative study with PC providers to evaluate the acceptability and perceived utility of the intervention.

Stage 1: Intervention development

The development of the proposed intervention involves:

1. Qualitative study with PC providers: the investigators will conduct three semi-structured interviews and four focus groups with PC doctors, nurses, and admin staff (n=36) to examine the acceptability and perceived utility of the proposed intervention, and to identify potential barriers towards wider implementation.
2. Translation and cross-cultural adaptation of the PREOS-PC instrument[8] into the Spanish context. The translation process, based on "state of the art" methods[9], will consist in forward and back translation by four independent translators, followed by cognitive interviews with eight to ten participants (diverse in terms of age, sex, and educational attainment) using the "think aloud" method [10] to ensure the translated version of the questionnaire is easy to understand and complete. The cross-cultural adaptation will be carried out using an expert consultation process involving five to seven national experts in PC patient safety.
3. Development of the intervention elements: the investigators will design the Feedback Report based on findings from previous studies[11-15] and from the qualitative study with PC providers above described. The Feedback Report will show the results of the Spanish PREOS-PC questionnaire specific for each PC centre. It will provide benchmarking data - i.e., practices will be able to see their individual scores compared to the average scores of the rest of participating practices. To facilitate the design of action plans to address the potential safety issues identified in the Feedback Report, the investigators will also produce a guidance document including a number of recommendations, good practices and materials to improve patient safety in PC, which will be identified as a result of a literature review of academic publications and key resources provided by national and international institutions, including the World Health Organization[16], the European Union Network for Patient Safety and Quality of Care (PaSQ Joint Action[17]), the Agency for healthcare research and quality[18], and the LINNEAUS EuroPC (Primary Care) collaboration[19], among others. The investigators will also produce a registry form to help PC centres register and monitor progress of the planned actions to address the safety problems identified. The intervention materials will also include information to increase PC providers´ awareness of the usefulness of patient elicited information as a strategy to identify potential safety problems and design strategies to address them.
4. Development of an online tool: the investigators will develop a bespoke online tool to allow the electronic administration of the PREOS-PC questionnaire to patients using tablet-computers. The data collected will be transferred to a database stored in a virtual server. Once all data has been collected from all participating patients in each PC centre, the tool will automatically generate and send the Feedback Reports to each of the participating centres. The tool will also be used to collect data from the healthcare professionals participating in the trial, which will be stored in a separate database. PC professionals will have password protected authentication to access to the provider questionnaire and to access to the Feedback Report.

Stage 2: Piloting the intervention, qualitative study and refining the intervention

Piloting the intervention will involve:

1. Feasibility study: the investigators will pilot the intervention in a three-month, one-arm (pre-post) feasibility trial. This will allow us to estimate the follow-up rate for the main trial; test the collection of the planned primary and secondary outcome data; the willingness of PC centres, providers and patients to participate; and the trial procedures. It will also allow us to examine the psychometric properties (floor and ceiling effects, internal consistency (calculating inter-item correlations[20] and Cronbach´s α[21]), and construct validity (confirmatory factor analysis)) of the Spanish PREOS-PC, and introduce final changes in the instrument if needed.

   Participants will include PC centres, providers and patients.

   Sample size: assuming an average of 26 healthcare professionals per centre, recruiting ten centres will result in approximately 260 professionals taking part in the feasibility trial. With 260 healthcare professionals, this feasibility study would allow us to detect 80% follow up rate within 95% confidence intervals of 75.1% to 84.8%. With 500 patients (50 per centre), the study is powered to detect a patient response rate to the questionnaire of 75% within 95% confidence intervals of 71.2% to 78.8%. 500 participants are sufficient to perform factor analyses and the rest of analyses planned for the evaluation of the psychometric properties of the Spanish PREOS-PC.

   Recruitment: the investigators will recruit 10 PC centres from the Balearic Islands diverse in terms of list size, deprivation, and rurality. The investigators will recruit patients, who will be approached in the waiting room by a research assistant and invited to complete the Spanish PREOS-PC.

   Statistical analysis. The investigators will calculate the overall provider follow-up rate as the proportion of healthcare providers that successfully complete the Spanish Medical Office Survey on Patient Safety Culture (MOSPSC)[22] at baseline and at three months post-intervention. The investigators will also calculate the follow-up rate by type of healthcare provider (nurse, doctor, social worker, administrative, etc.). Response rate to the patient questionnaire will also be calculated. This will include total response rate and response rate by centre and patient characteristics (age and gender).
2. Embedded qualitative study: after the intervention period the investigators will conduct semi-structured qualitative interviews with 20 healthcare professionals. They will be purposefully selected to ensure variation in terms of professional roles. Thematic analysis [23] will be used to explore the acceptability and perceived utility of the intervention, as well as possible suggestions to improve the intervention delivery or content.
3. Refining the intervention: Results from the feasibility trial will be used to inform the potential refinements of the online tool to collect data and generate the Feedback Reports, also about the intervention as well as the trials procedures. The investigators will carry out an explicit process to decide the final intervention content, including a systematic appraisal of the trial processes (both quantitative and qualitative data) and proposals for solutions to identified problems.

Stage 3: Evaluating the acceptability, perceived utility and effectiveness of the intervention

The evaluation of the intervention will involve:

1. Cluster randomized controlled trial: the investigators will conduct a multi-centre, 12 month, two-arm, two-level cluster randomized controlled trial (PC professionals within PC centres; with randomization at the centre level in a 1:1 ratio). A cluster randomised trial is proposed to avoid the risk of contamination across professionals working in the same centre. 24 PC centres will be allocated to the control group and 24 to the intervention group. PC centres in the intervention group will receive the intervention described above. Centres in the control group will not receive any intervention during the study period but will receive the Feedback Reports at the end of the study.

   Randomization: Randomization will be done using a fully validated randomisation algorithm. Allocation will be carried out using a non-deterministic minimisation algorithm to ensure PC centres are balanced for important characteristics (including region, deprivation, and list size) and baseline measures.

   Participants: staff working and patients registered in the included PC centres.

   Sample size: The sample size calculation for this trial is based on its main outcome measure - the Spanish version of the MOSPSC, which ranges from 1-5. Assuming an average of 26 professionals per centre, approximately 1,248 professionals will take part in the study (624 in the intervention and 624 in the control group). Assuming a follow-up rate of 80%, the investigators will have complete data from approximately 998 professionals. Taking into account the cluster design, and using a conservative estimation of intra-class correlation of 0.1, this sample size will allow us to detect at least a 0.3 difference in effect size (with 80% power and a significance level of 5%). This would approximately correspond to a difference of 0.8 points in the index (assuming standard deviation of 2.3 from a previous study) [24]. The investigators will recruit 75 patients per centre (3,600 in total) because, according to the psychometric study of the original version of PREOS-PC[8], that is the number of questionnaires needed to achieve a 0.7 reliability of scale scores at the centre level. A more precise sample size calculation will be possible after the completion of the feasibility trial above described.

   Recruitment and training of PC centres: The investigators will recruit 48 PC centres from Balearic Islands and other regions in Spain. Centres will be recruited through scientific societies and key informants. Centres will be purposefully selected in order to ensure variation in terms of list size, rurality and levels of deprivation. Centres will be asked to consent as a unit, with all professionals being willing to participate. Consent will also be taken from patients invited to complete the patient survey.

   Data collection: Data will be collected at baseline and 12 months post-intervention (i.e. 12 months after the Feedback Reports are sent to the centres). The investigators will monitor the progress of the intervention in all the centres. Data from patients will include patient reported experiences and outcomes of patient safety in PC (measured with PREOS-PC) and patient sociodemographic characteristics. Data from healthcare professionals will be collected through online questionnaires and will include the perceived safety climate (measured with the Spanish MOSPSC), and sociodemographic and occupational characteristics. Data from centres will include rate of avoidable hospitalizations in the previous 12 months (which will be extracted from electronic medical records), and centre characteristics (rurality, list size, number of healthcare professionals, and deprivation index).

   Statistical analyses: Baseline variables will be presented by randomised group using frequencies (with percentages) for binary and categorical variables and means (and standard deviations) or medians (interquartile range) for continuous variables. The results from the trial will be presented as comparative summary statistics (difference in proportions or means) with 95% confidence intervals. The primary outcome will be analysed using a hierarchical model, with individuals (PC professionals) nested within PC centres in an analysis of covariance adjusted for minimisation factors. All analyses will be carried out on the basis of intention-to-treat (ITT).
2. Qualitative study with PC providers (within trial qualitative evaluation): An embedded qualitative study will be carried out to understand the way the intervention is perceived among PC professionals in terms of acceptability, perceived utility and implementation barriers (including any unintended consequences). Around 30 PC professionals in the intervention centres will be invited to take part in an interview at the end of the trial. The investigators will use purposeful sampling in order to ensure variation in terms of type of PC professionals (doctors, nurses, administrative staff, etc.) and of centres (region, rurality, deprivation, list size). Interviews will take place in the centres or telephonically. Thematic analysis[23] will be used to identify recurrent themes and subthemes common to interviewees working in centres.

ELIGIBILITY:
Inclusion Criteria:

* patients who to have visited their PC centre at least once in the previous 12 months.
* have to be able to speak Spanish

Exclusion Criteria:

* overt psychosis/critically ill/altered mental status
* inability to provide written informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1248 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in the Patient Safety Climate Synthetic Index | At pre-intervention and after 12 months follow-up
  Measured with the Spanish version of the Medical Office Survey on Patient Safety Culture (MOSPSC) at the PC professional level. This scale measures safety culture of the primary health centres.

SECONDARY OUTCOMES:
Patient Reported Experiences and Outcomes of Safety in Primary Care (PREOS-PC): Centre Activation | At pre-intervention and after 12 months follow-up
  Patient-Reported Patient Safety questionnaire measures the patient safety experiences in Primary Care settings. The following scales from the Spanish PREOS-PC will be used (the range is from 0 to 100. Higher scores indicate better results)
  • Centre Activation (11 items; Cronbach's α of the original version=0.89). Average score of the scale.
  For each scale, PC centre level scores will be calculated as the mean score from patients registered in the PC centre. Patient scores will be calculated as the percentage of the maximum score achievable on all items.
Patient Reported Experiences and Outcomes of Safety in Primary Care (PREOS-PC): Patient Activation | At pre-intervention and after 12 months follow-up
  Patient-Reported Patient Safety questionnaire measures the patient safety experiences in Primary Care settings. The following scales from the Spanish PREOS-PC will be used (for each scale the range is from 0 to 100. Higher scores indicate better results)
  • Patient Activation (2 items; α=0.80). Average score of the scale.
  For each scale, PC centre level scores will be calculated as the mean score from patients registered in the PC centre. Patient scores will be calculated as the percentage of the maximum score achievable on all items.
Patient Reported Experiences and Outcomes of Safety in Primary Care (PREOS-PC): Experiences of Safety Problems | At pre-intervention and after 12 months follow-up
  Patient-Reported Patient Safety questionnaire measures the patient safety experiences in Primary Care settings. The following scales from the Spanish PREOS-PC will be used (for each scale the range is from 0 to 100. Higher scores indicate better results)
  • Experiences of Safety Problems (12 items; α= 0.75). Percentage of safety problems.
  For each scale, PC centre level scores will be calculated as the mean score from patients registered in the PC centre. Patient scores will be calculated as the percentage of the maximum score achievable on all items.
Patient Reported Experiences and Outcomes of Safety in Primary Care (PREOS-PC): Harm | At pre-intervention and after 12 months follow-up
  Patient-Reported Patient Safety questionnaire measures the patient safety experiences in Primary Care settings. The following scales from the Spanish PREOS-PC will be used (for each scale the range is from 0 to 100. Higher scores indicate better results)
  • Harm (5 items; α=0.96). Average score of the scale.
  For each scale, PC centre level scores will be calculated as the mean score from patients registered in the PC centre. Patient scores will be calculated as the percentage of the maximum score achievable on all items.
Patient Reported Experiences and Outcomes of Safety in Primary Care (PREOS-PC): Overall rating of patient safety | At pre-intervention and after 12 months follow-up
  Patient-Reported Patient Safety questionnaire measures the patient safety experiences in Primary Care settings. The following scales from the Spanish PREOS-PC will be used (for each scale the range is from 0 to 100. Higher scores indicate better results)
  • Overall rating of patient safety (1 item). Average score of the scale.
  For each scale, PC centre level scores will be calculated as the mean score from patients registered in the PC centre. Patient scores will be calculated as the percentage of the maximum score achievable on all items.
Rate of avoidable hospitalizations | At pre-intervention and after 12 months follow-up
  Calculated as the number of avoidable hospitalizations per 1,000 patients in the last 12 months. Data on avoidable hospitalizations will be extracted from electronic medical records using available International Classification Diseases (CIE-9) codes

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio Ricci-Cabello, PhD, Principal Investigator — Institut d'Investigació Sanitària de les Illes Balears
Locations (1):
- Ignacio Ricci-Cabello, Palma de Mallorca, Balearic Islands, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Institute of Medicine (US) Committee on Quality of Health Care in America; Kohn LT, Corrigan JM, Donaldson MS, editors. To Err is Human: Building a Safer Health System. Washington (DC): National Academies Press (US); 2000. Available from http://www.ncbi.nlm.nih.gov/books/NBK225182/ PMID 25077248
- [Background] Woods DM, Thomas EJ, Holl JL, Weiss KB, Brennan TA. Ambulatory care adverse events and preventable adverse events leading to a hospital admission. Qual Saf Health Care. 2007 Apr;16(2):127-31. doi: 10.1136/qshc.2006.021147. PMID 17403759
- [Background] Green LA, Fryer GE Jr, Yawn BP, Lanier D, Dovey SM. The ecology of medical care revisited. N Engl J Med. 2001 Jun 28;344(26):2021-5. doi: 10.1056/NEJM200106283442611. No abstract available. PMID 11430334
- [Background] Aranaz-Andres JM, Aibar C, Limon R, Mira JJ, Vitaller J, Agra Y, Terol E. A study of the prevalence of adverse events in primary healthcare in Spain. Eur J Public Health. 2012 Dec;22(6):921-5. doi: 10.1093/eurpub/ckr168. Epub 2011 Nov 29. PMID 23180803
- [Background] Kluger, A.N. and A. DeNisi, The effects of feedback interventions on performance: a historical review, a meta-analysis, and a preliminary feedback intervention theory. Psychological bulletin, 1996. 119(2): p. 254.
- [Background] Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M. Developing and evaluating complex interventions: the new Medical Research Council guidance. Int J Nurs Stud. 2013 May;50(5):587-92. doi: 10.1016/j.ijnurstu.2012.09.010. Epub 2012 Nov 15. No abstract available. PMID 23159157
- [Background] Ricci-Cabello I, Avery AJ, Reeves D, Kadam UT, Valderas JM. Measuring Patient Safety in Primary Care: The Development and Validation of the "Patient Reported Experiences and Outcomes of Safety in Primary Care" (PREOS-PC). Ann Fam Med. 2016 May;14(3):253-61. doi: 10.1370/afm.1935. PMID 27184996
- [Background] Wild D, Grove A, Martin M, Eremenco S, McElroy S, Verjee-Lorenz A, Erikson P; ISPOR Task Force for Translation and Cultural Adaptation. Principles of Good Practice for the Translation and Cultural Adaptation Process for Patient-Reported Outcomes (PRO) Measures: report of the ISPOR Task Force for Translation and Cultural Adaptation. Value Health. 2005 Mar-Apr;8(2):94-104. doi: 10.1111/j.1524-4733.2005.04054.x. PMID 15804318
- [Background] Someren, Maarten & Barnard, Yvonne & Sandberg, Jacobijn. (1994). The Think Aloud Method - A Practical Guide to Modelling Cognitive Processes.
- [Background] Boyce MB, Browne JP. Does providing feedback on patient-reported outcomes to healthcare professionals result in better outcomes for patients? A systematic review. Qual Life Res. 2013 Nov;22(9):2265-78. doi: 10.1007/s11136-013-0390-0. Epub 2013 Mar 17. PMID 23504544
- [Background] Kasbauer S, Cooper R, Kelly L, King J. Barriers and facilitators of a near real-time feedback approach for measuring patient experiences of hospital care. Health Policy Technol. 2017 Mar;6(1):51-58. doi: 10.1016/j.hlpt.2016.09.003. PMID 28367401
- [Background] Lawton R, O'Hara JK, Sheard L, Armitage G, Cocks K, Buckley H, Corbacho B, Reynolds C, Marsh C, Moore S, Watt I, Wright J. Can patient involvement improve patient safety? A cluster randomised control trial of the Patient Reporting and Action for a Safe Environment (PRASE) intervention. BMJ Qual Saf. 2017 Aug;26(8):622-631. doi: 10.1136/bmjqs-2016-005570. Epub 2017 Feb 3. PMID 28159854
- [Background] Porter I, Goncalves-Bradley D, Ricci-Cabello I, Gibbons C, Gangannagaripalli J, Fitzpatrick R, Black N, Greenhalgh J, Valderas JM. Framework and guidance for implementing patient-reported outcomes in clinical practice: evidence, challenges and opportunities. J Comp Eff Res. 2016 Aug;5(5):507-19. doi: 10.2217/cer-2015-0014. Epub 2016 Jul 18. PMID 27427277
- [Background] Greenhalgh J, Dalkin S, Gooding K, Gibbons E, Wright J, Meads D, Black N, Valderas JM, Pawson R. Functionality and feedback: a realist synthesis of the collation, interpretation and utilisation of patient-reported outcome measures data to improve patient care. Southampton (UK): NIHR Journals Library; 2017 Jan. Available from http://www.ncbi.nlm.nih.gov/books/NBK409450/ PMID 28121094
- [Background] Nunnally, J.C. and I.H. Bernstein, Psychometric theory. Vol. 226. 1967: McGraw-Hill New York.
- [Background] Silvestre-Busto C, Torijano-Casalengua ML, Olivera-Canadas G, Astier-Pena MP, Maderuelo-Fernandez JA, Rubio-Aguado EA. [Adaptation of the Medical Office Survey on Patient Safety Culture (MOSPSC) tool]. Rev Calid Asist. 2015 Jan-Feb;30(1):24-30. doi: 10.1016/j.cali.2014.12.006. Epub 2015 Feb 7. Spanish. PMID 25659444
- [Background] Guest, G., K.M. MacQueen, and E.E. Namey, Applied thematic analysis. 2011: sage.
- [Background] Ricci-Cabello I, Marsden KS, Avery AJ, Bell BG, Kadam UT, Reeves D, Slight SP, Perryman K, Barnett J, Litchfield I, Thomas S, Campbell SM, Doos L, Esmail A, Valderas JM. Patients' evaluations of patient safety in English general practices: a cross-sectional study. Br J Gen Pract. 2017 Jul;67(660):e474-e482. doi: 10.3399/bjgp17X691085. Epub 2017 Jun 5. PMID 28583945
- [Derived] Fiol-deRoque MA, Valderas JM, Serrano-Ripoll MJ, Gens-Barbara M, Martin-Lujan F, Sanchez-Freire E, Montano JJ, Mira-Martinez S, Pastor-Moreno G, Zamanillo-Campos R, Riera-Serra P, Ricci-Cabello I. Evaluating SinergiAPS, an intervention based on patient feedback to improve patient safety in primary care: a cluster randomized trial. BMC Med. 2025 Apr 7;23(1):202. doi: 10.1186/s12916-025-04029-7. PMID 40189506
- [Derived] Serrano-Ripoll MJ, Ripoll J, Llobera J, Valderas JM, Pastor-Moreno G, Olry de Labry Lima A, Ricci-Cabello I. Development and evaluation of an intervention based on the provision of patient feedback to improve patient safety in Spanish primary healthcare centres: study protocol. BMJ Open. 2019 Dec 23;9(12):e031367. doi: 10.1136/bmjopen-2019-031367. PMID 31874872
- See also: Related Info — https://www.wiley.com/en-es/Patient+Safety,+2nd+Edition-p-9781405192217
- See also: Agency for Healthcare Research and Quality — http://www.ahrq.gov.
- See also: Learning from International Networks about Errors and Understanding Safety in Primary Care — https://cordis.europa.eu/project/rcn/90964/reporting/en